CLINICAL TRIAL: NCT00562887
Title: A Phase 2B, Multi-Center, Randomized, Double-blind, Parallel Group, Placebo-controlled, Dose Ranging Study Comparing the Efficacy, Safety and Pharmacokinetics of Intravenous Infusions of ABT-874 vs. Placebo in Subjects With Moderately to Severely Active Crohn's Disease.
Brief Title: Dose Ranging Study Comparing the Efficacy, Safety and Pharmacokinetics of Intravenous Infusions of ABT-874 vs Placebo in Subjects With Active Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-222; 2008-004919-36 (Registry Identifier: EudraCT)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — briakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Biological: Placebo
- 400 mg (Experimental)
  Interventions: Biological: ABT-874
- 700mg (Experimental)
  Interventions: Biological: ABT-874

INTERVENTIONS:
Biological: Placebo — every 4 weeks, IV
  Arms: 1
Biological: ABT-874 — 400 mg IV every 4 weeks
  Arms: 400 mg
Biological: ABT-874 — 700 mg IV every 4 weeks
  Arms: 700mg

SUMMARY:
To compare the efficacy, safety and pharmacokinetics of ABT-874 to placebo in subjects who have moderately to severely active Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease for greater than 4 months confirmed by endoscopy or radiologic evaluation.
* CDAI score of >= 220 and <= 450 at Week 0.
* Males and females >= 18 years and < 75 years of age at the Screening visit.
* Judged to be in generally good health as determined by the Investigator.

Exclusion Criteria:

* Current diagnosis of the colitis other than Crohn's disease.
* Symptomatic known strictures.
* Surgical bowel resections within the past 6 months or is planning any resection at any time point while enrolled in the study.
* Ostomy or ileoanal pouch. (Subjects with a previous ileo-rectal anastomosis are not excluded).
* Short bowel syndrome as determined by the investigator.
* Infection or risk factors for severe infections.
* Females who are pregnant or considering becoming pregnant during the study, or breast-feeding.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical remission, defined as CDAI score of <150 points | Week 6

SECONDARY OUTCOMES:
Patient reported outcomes, clinical response indicators, safety parameters | Weeks 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Carcereri, MD, Study Director — Abbott
Locations (61):
- United States (36):
  - Site Ref # / Investigator 6792, Orange, California
  - Site Ref # / Investigator 6643, San Diego, California
  - Site Ref # / Investigator 6670, Hamden, Connecticut
  - Site Ref # / Investigator 6694, Gainesville, Florida
  - Site Ref # / Investigator 6794, Jacksonville, Florida
  - Site Ref # / Investigator 6687, Winter Park, Florida
  - Site Ref # / Investigator 6667, Zephyrhills, Florida
  - Site Ref # / Investigator 6691, Atlanta, Georgia
  - Site Ref # / Investigator 6642, Atlanta, Georgia
  - Site Ref # / Investigator 8797, Macon, Georgia
  - Site Ref # / Investigator 6925, Baton Rouge, Louisiana
  - Site Ref # / Investigator 6865, Chevy Chase, Maryland
  - Site Ref # / Investigator 10202, Towson, Maryland
  - Site Ref # / Investigator 6866, Rochester, Minnesota
  - Site Ref # / Investigator 6778, Mexico, Missouri
  - Site Ref # / Investigator 7048, St Louis, Missouri
  - Site Ref # / Investigator 7952, Las Vegas, Nevada
  - Site Ref # / Investigator 6647, Cedar Knolls, New Jersey
  - Site Ref # / Investigator 6689, Great Neck, New York
  - Site Ref # / Investigator 6652, Lake Success, New York
  - Site Ref # / Investigator 7047, New York, New York
  - Site Ref # / Investigator 6693, Asheville, North Carolina
  - Site Ref # / Investigator 6785, Charlotte, North Carolina
  - Site Ref # / Investigator 9070, Morgantown, North Carolina
  - Site Ref # / Investigator 6651, Raleigh, North Carolina
  - Site Ref # / Investigator 6665, Beachwood, Ohio
  - Site Ref # / Investigator 6690, Cincinnati, Ohio
  - Site Ref # / Investigator 6786, Portland, Oregon
  - Site Ref # / Investigator 7004, Germantown, Tennessee
  - Site Ref # / Investigator 6648, Nashville, Tennessee
  - Site Ref # / Investigator 6793, Nashville, Tennessee
  - Site Ref # / Investigator 7054, Nashville, Tennessee
  - Site Ref # / Investigator 8357, Round Rock, Texas
  - Site Ref # / Investigator 6688, Ogden, Utah
  - Site Ref # / Investigator 9115, Chesapeake, Virginia
  - Site Ref # / Investigator 6674, Seattle, Washington
- Site Ref # / Investigator 16983, Box Hill, Victoria, Australia
- Site Ref # / Investigator 16225, Vienna, Austria
- Belgium (2):
  - Site Ref # / Investigator 16230, Bonheiden
  - Site Ref # / Investigator 16231, Leuven
- Canada (16):
  - Site Ref # / Investigator 9422, Calgary, Alberta
  - Site Ref # / Investigator 14042, Edmonton, Alberta
  - Site Ref # / Investigator 7610, Vancouver, British Columbia
  - Site Ref # / Investigator 8206, Winnipeg, Manitoba
  - Site Ref # / Investigator 7634, St. John's, Newfoundland and Labrador
  - Site Ref # / Investigator 7596, Halifax, Nova Scotia
  - Site Ref # / Investigator 7630, Truro, Nova Scotia
  - Site Ref # / Investigator 7641, Hamilton, Ontario
  - Site Ref # / Investigator 10681, London, Ontario
  - Site Ref # / Investigator 17901, Toronto, Ontario
  - Site Ref # / Investigator 7629, Montreal, Quebec
  - Site Ref # / Investigator 14702, Montreal, Quebec
  - Site Ref # / Investigator 15061, Montreal, Quebec
  - Site Ref # / Investigator 17881, Québec, Quebec
  - Site Ref # / Investigator 7642, Saskatoon, Saskatchewan
  - Site Ref # / Investigator 14821, Saskatoon, Saskatchewan
- Denmark (3):
  - Site Ref # / Investigator 16985, Herlev
  - Site Ref # / Investigator 16235, Hvivdovre
  - Site Ref # / Investigator 16234, Odense C
- Puerto Rico (2):
  - Site Ref # / Investigator 10961, Ponce
  - Site Ref # / Investigator 16801, San Juan